CLINICAL TRIAL: NCT06423794
Title: A Phase 2, Multicenter, Open-Label Extension Study to Assess the Long-Term Safety and Tolerability of BHV-7000 in Treatment of Bipolar I Disorder
Brief Title: BHV-7000 Open-Label Extension Bipolar Mania Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business Decision
Sponsor: Biohaven Therapeutics Ltd. (Industry)
Responsible Party: Sponsor
Organization: Biohaven Pharmaceuticals, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BHV7000-202
Record Dates: First submitted 2024-05-16; First posted 2024-05-21 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Bipolar Disorder
Keywords: bipolar; mania; manic episode; manic state; bipolar disorder type 1; manic depressive; manic bipolar; mixed features; mixed episode; mixed mania; bipolar episode; bipolar disorder
MeSH Terms: conditions — Bipolar Disorder; Mania

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BHV-7000 (Experimental)
  Interventions: Drug: BHV-7000

INTERVENTIONS:
Drug: BHV-7000 — BHV-7000 75 mg taken once daily

SUMMARY:
The purpose of this study is to evaluate the long-term safety and tolerability of BHV-7000 in subjects with bipolar I disorder.

ELIGIBILITY:
Key Inclusion Criteria:

1. Subjects must have successfully completed the parent study, BHV7000-204.
2. WOCBP must have a negative urine pregnancy test at Baseline visit.
3. WOCBP must not be breastfeeding or lactating at Baseline visit or any point in the study.

Key Exclusion Criteria:

1. Any medical condition, based on the judgement of the Investigator, that would confound the ability to adequately assess safety and efficacy outcome measures.
2. Subjects who, in the opinion of the Investigator, will not be able to adhere to the Schedule of Assessments and/or may have difficulties complying with the treatment regimen over an extended duration of a long-term, outpatient study.
3. Investigator deems subject at imminent risk of danger to others or themself.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2024-06-24 (Actual); Primary Completion 2025-04-25 (Actual); Study Completion 2025-04-25 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Clinically Significant Laboratory Abnormalities | Up to 52 weeks
  To assess the safety and tolerability of BHV-7000. This objective will be measured by assessing the number of unique subjects with grade 3 or 4 laboratory abnormalities.
Number of Participants With Serious AEs (SAEs), AEs Leading to Study Drug Discontinuation, and AEs judged to be related to study medication | Up to 52 weeks
  To assess the safety and tolerability of BHV-7000. This objective will be measured by assessing the number of unique subjects with SAEs, AEs leading to discontinuation, AEs judged to be related to study medication that are observed during the Double-blind Treatment Phase (21 days).
Number of Participants With Vital Sign Abnormalities | Up to 52 weeks
Number of Participants With Electrocardiogram (ECG) Abnormalities specific to QTc elevation | Up to 52 weeks

CONTACTS AND LOCATIONS:
Locations (32):
- United States (32):
  - Pillar Clinical Research, LLC, Bentonville, Arkansas
  - WIRG, Little Rock, Arkansas
  - WRN, Rogers, Arkansas
  - Advanced Research Center, Inc., Anaheim, California
  - CIT LA, Bellflower, California
  - ProScience Research Group, Culver City, California
  - Cenexel CNS, Garden Grove, California
  - Synergy San Diego, Lemon Grove, California
  - NRC Research Institute, Orange, California
  - CIT IE, Riverside, California
  - Cenexel CNS, Torrance, California
  - Segal Trials - Larkin Behavioral Health Services-Inpatient & Early Phase Site, Hollywood, Florida
  - Cenexel - RCA, Hollywood, Florida
  - LCC Medical Research Inst, Miami, Florida
  - Floridian Neuroscience Institute, Miami Lakes, Florida
  - Segal Trials - Miami Lakes Medical Research-Inpatient & Early Phase Site, Miami Lakes, Florida
  - Neuroscience Research Institute, West Palm Beach, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - CenExel iResearch, LLC, Decatur, Georgia
  - CenExel iResearch, LLC, Savannah, Georgia
  - Uptown Research Institute, Chicago, Illinois
  - Pillar Clinical Research, Chicago, Illinois
  - CBH Health, Gaithersburg, Maryland
  - Precise Clinical Research, Flowood, Mississippi
  - Arch Clinical Trials, St Louis, Missouri
  - Hassman Research Institute, Marlton, New Jersey
  - RBA, Staten Island, New York
  - Midwest Clinical Research Center, Dayton, Ohio
  - NBCR, North Canton, Ohio
  - Community Clinical Research, Inc., Austin, Texas
  - InSite Clinical Research, LLC, DeSoto, Texas
  - Pillar Clinical Research, LLC, Richardson, Texas